CLINICAL TRIAL: NCT01134549
Title: A Double-Blind, Randomized, Placebo-Controlled, Rising Single Intravenous Dose Study to Assess the Safety, Tolerability and Pharmacokinetics of KAI-4169 in Healthy Male Volunteers
Brief Title: Safety, Tolerability and Pharmacokinetics of Etelcalcetide in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KAI Pharmaceuticals (Industry)
Collaborators: Nucleus Network Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAI-4169-001; 20130107 (Other: Amgen, Inc)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-02

CONDITIONS: Hyperparathyroidism, Secondary
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — etelcalcetide hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received a single dose of placebo intravenous injection.
  Interventions: Drug: Placebo
- Etelcalcetide (Experimental): Participants received a single dose of etelcalcetide intravenous injection; the starting dose was 0.5 mg.
  Interventions: Drug: Etelcalcetide

INTERVENTIONS:
Drug: Etelcalcetide — Administered as a single intravenous (IV) injection
  Other Names: KAI-4169; AMG 416; Parsabiv™
  Arms: Etelcalcetide
Drug: Placebo — Administered as a single intravenous (IV) injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to characterize the safety and tolerability of etelcalcetide in healthy young males.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 45 years of age who have provided written informed consent
* Subject is judged to be in good health based on medical history, physical examination, and routine laboratory tests

Exclusion Criteria:

* History or presence of any significant acute or chronic illness (e.g., cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, or neurologic disease) according to the investigator
* History of any ongoing medical condition requiring treatment with prescription medication
* History of asthma, severe allergies including skin reactions or prior anaphylactic type reactions
* Clinically significant abnormalities on screening clinical examination or laboratory safety tests
* History of drug or alcohol abuse

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-06-09; Primary Completion 2010-07-31 (Actual); Study Completion 2010-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M D, Study Director — Amgen
Locations (1):
- Melbourne, Victoria, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one clinical center in Australia.
Pre-assignment Details: The study included 4 cohorts: 0.5 mg, 2 mg, 5 mg and 10 mg. Eight participants were enrolled into each cohort and were randomized 6:2 to receive etelcalcetide or placebo.
Groups:
- Pooled Placebo: Participants received a single dose of placebo administered by intravenous injection.
- Etelcalcetide 0.5 mg: Participants received a single dose of 0.5 mg etelcalcetide administered by intravenous injection.
- Etelcalcetide 2 mg: Participants received a single dose of 2 mg etelcalcetide administered by intravenous injection.
- Etelcalcetide 5 mg: Participants received a single dose of 5 mg etelcalcetide administered by intravenous injection.
- Etelcalcetide 10 mg: Participants received a single dose of 10 mg etelcalcetide administered by intravenous injection.
Period: Overall Study
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Started | 8 | 6 | 6 | 6 | 6
Completed | 8 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Total
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (3.5) | 27.8 (8.9) | 26.8 (4.9) | 24.2 (4.4) | 26.0 (6.2) | 25.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 6 | 6 | 6 | 6 | 32
Race [Count of Participants; unit: Participants]
  White | 6 | 4 | 6 | 3 | 4 | 23
  Asian | 2 | 2 | 0 | 2 | 2 | 8
  Other | 0 | 0 | 0 | 1 | 0 | 1
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 8 | 6 | 5 | 6 | 6 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: From the first dose of study drug through 7 days.
Population: The modified intent-to-treat (MITT) population consisted of all participants who were randomized and received study medication.
Measure: Number; unit: participants
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
participants
  Any adverse event | 2 | 0 | 1 | 2 | 2
  Serious adverse events | 0 | 0 | 0 | 0 | 0
  Withdrawals due to adverse events | 0 | 0 | 0 | 0 | 0
  Treatment-related adverse events | 0 | 0 | 1 | 1 | 1
  Deaths | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Percent Change From Baseline in Serum Parathyroid Hormone
Time Frame: Baseline and 10 minutes, 30 minutes, 1 hour, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 36, 42 and 48 hours post-dose
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
percent change
  10 Minutes | 4.57 (15.42) | -20.58 (4.25) | -45.09 (9.31) | -59.38 (8.89) | -63.31 (8.11)
  30 Minutes | -3.52 (16.29) | -21.74 (9.55) | -55.42 (4.31) | -69.00 (7.02) | -72.56 (6.33)
  1 Hour | 1.11 (12.85) | -18.71 (11.68) | -47.16 (7.94) | -67.72 (10.84) | -73.29 (6.97)
  3 Hours | 1.76 (26.67) | -5.95 (7.62) | -39.87 (10.87) | -62.56 (13.30) | -69.70 (7.62)
  6 Hours | -2.57 (30.28) | 7.01 (10.64) | -41.56 (12.03) | -60.87 (13.41) | -66.68 (10.41)
  9 Hours | 19.87 (25.16) | 46.50 (27.97) | 12.54 (40.52) | -40.79 (15.91) | -54.43 (12.97)
  12 Hours | 30.49 (28.14) | 8.07 (17.54) | 5.04 (27.93) | -24.05 (13.94) | -40.28 (19.35)
  15 Hours | 31.97 (25.22) | 4.17 (19.38) | 20.06 (39.27) | -2.33 (21.12) | -24.31 (17.06)
  18 Hours | 27.21 (15.21) | -6.22 (11.89) | 25.91 (28.39) | 2.19 (20.72) | -15.78 (13.66)
  21 Hours | 9.65 (16.08) | -0.67 (20.04) | 22.04 (16.74) | -2.10 (25.36) | -4.02 (19.11)
  24 Hours | -9.50 (16.20) | -1.72 (22.40) | -14.65 (13.43) | -19.25 (17.66) | -18.34 (15.17)
  27 Hours | -21.56 (11.39) | -27.97 (10.32) | -34.76 (13.58) | -49.48 (12.23) | -37.15 (18.99)
  30 Hours | 10.58 (15.51) | -8.19 (14.90) | 1.21 (21.70) | -11.15 (23.59) | -25.32 (12.63)
  36 Hours | 25.24 (20.51) | 18.19 (25.35) | 20.63 (34.27) | 17.61 (37.53) | 1.08 (27.77)
  42 Hours | 6.15 (26.47) | 3.28 (11.15) | 1.49 (23.88) | -19.21 (20.33) | -29.37 (21.78)
  48 Hours | -13.90 (15.92) | -10.39 (12.66) | -4.86 (26.04) | -24.02 (15.00) | -10.84 (20.60)

3. Secondary Outcome: Percent Change From Baseline in Plasma Ionized Calcium
Time Frame: Baseline and 10 minutes, 30 minutes, 1 hour, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 36, 42 and 48 hours post-dose
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
percent change
  10 Minutes | -1.48 (3.55) | 0.98 (2.79) | -3.94 (2.33) | -5.30 (2.13) | -2.47 (2.79)
  30 Minutes | -1.27 (3.67) | -0.51 (3.54) | -2.46 (3.20) | -6.87 (2.06) | 1.18 (2.92)
  1 Hour | -1.15 (4.62) | 1.15 (3.08) | -4.50 (2.65) | -4.12 (2.08) | -3.27 (1.52)
  3 Hours | -1.72 (4.85) | 0.73 (1.40) | -5.86 (2.52) | -6.65 (2.31) | -1.83 (4.07)
  6 Hours | -1.79 (3.32) | -1.36 (2.66) | -4.88 (2.58) | -9.95 (1.91) | -2.84 (2.67)
  9 Hours | -4.68 (3.76) | -3.39 (5.00) | -9.51 (5.40) | -16.45 (2.55) | -9.54 (5.32)
  12 Hours | -7.14 (3.93) | -2.83 (3.22) | -9.54 (2.17) | -15.27 (1.49) | -14.92 (5.47)
  15 Hours | -3.71 (4.25) | -2.53 (2.98) | -10.41 (1.32) | -15.38 (3.05) | -11.74 (4.08)
  18 Hours | -3.38 (4.24) | -1.62 (5.07) | -9.00 (1.18) | -14.33 (2.31) | -12.34 (3.27)
  21 Hours | -1.11 (3.56) | 3.90 (3.60) | -6.38 (1.74) | -13.97 (2.48) | -11.77 (1.85)
  24 Hours | -0.70 (4.64) | 3.77 (1.93) | -2.45 (1.95) | -11.83 (4.46) | -11.59 (4.49)
  27 Hours | -1.78 (4.12) | 2.62 (3.73) | -6.26 (2.74) | -7.71 (2.28) | -7.89 (1.46)
  30 Hours | 0.17 (4.11) | 2.51 (3.84) | -5.82 (2.06) | -9.65 (2.73) | -11.78 (5.66)
  36 Hours | -5.02 (5.40) | -3.28 (5.39) | -7.68 (3.35) | -13.69 (4.43) | -9.45 (3.11)
  42 Hours | -1.38 (3.56) | 0.55 (3.44) | 0.14 (1.32) | -5.92 (3.30) | -3.40 (3.07)
  48 Hours | 2.12 (4.24) | 2.17 (2.91) | -0.42 (1.83) | -6.22 (3.17) | -0.39 (2.85)

4. Secondary Outcome: Change From Baseline in Serum Total Calcium
Time Frame: Baseline and 10 minutes, 30 minutes, 1 hour, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 36, 42 and 48 hours post-dose
Population: Modified intent-to-treat population with available data at each time point
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
mmol/L
  10 Minutes: number analyzed (Participants) | 7 | 6 | 6 | 6 | 6
  10 Minutes | -0.019 (0.047) | -0.008 (0.081) | -0.022 (0.063) | -0.017 (0.053) | -0.030 (0.049)
  30 Minutes | -0.018 (0.036) | -0.008 (0.079) | -0.018 (0.062) | -0.023 (0.041) | -0.042 (0.037)
  1 Hour | -0.024 (0.039) | -0.033 (0.073) | -0.023 (0.056) | -0.017 (0.058) | -0.042 (0.026)
  3 Hours: number analyzed (Participants) | 7 | 6 | 6 | 6 | 6
  3 Hours | -0.001 (0.035) | -0.018 (0.074) | -0.017 (0.048) | -0.025 (0.066) | -0.050 (0.032)
  6 Hours: number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
  6 Hours | -0.024 (0.040) | -0.065 (0.090) | 0.008 (0.066) | -0.045 (0.058) | -0.138 (0.061)
  9 Hours: number analyzed (Participants) | 8 | 5 | 6 | 5 | 6
  9 Hours | -0.010 (0.041) | -0.122 (0.117) | -0.120 (0.218) | -0.126 (0.043) | -0.170 (0.065)
  12 Hours | -0.055 (0.038) | -0.058 (0.080) | -0.067 (0.024) | -0.203 (0.041) | -0.285 (0.079)
  15 Hours | -0.176 (0.324) | -0.075 (0.105) | -0.107 (0.039) | -0.243 (0.064) | -0.312 (0.056)
  18 Hours | -0.090 (0.074) | -0.030 (0.077) | -0.100 (0.027) | -0.217 (0.045) | -0.328 (0.075)
  21 Hours: number analyzed (Participants) | 8 | 6 | 6 | 5 | 6
  21 Hours | -0.058 (0.038) | -0.012 (0.113) | -0.090 (0.041) | -0.174 (0.040) | -0.285 (0.039)
  24 Hours: number analyzed (Participants) | 8 | 6 | 6 | 5 | 5
  24 Hours | -0.025 (0.030) | -0.040 (0.076) | -0.038 (0.061) | -0.200 (0.036) | -0.270 (0.072)
  27 Hours | 0.030 (0.037) | 0.020 (0.106) | 0.018 (0.080) | -0.070 (0.057) | -0.165 (0.058)
  30 Hours: number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
  30 Hours | -0.003 (0.036) | 0.025 (0.102) | -0.013 (0.063) | -0.165 (0.071) | -0.182 (0.057)
  36 Hours | -0.035 (0.035) | -0.002 (0.074) | -0.058 (0.084) | -0.143 (0.077) | -0.210 (0.040)
  42 Hours: number analyzed (Participants) | 8 | 6 | 6 | 5 | 6
  42 Hours | -0.009 (0.055) | -0.033 (0.085) | 0.002 (0.029) | -0.100 (0.021) | -0.120 (0.045)
  48 Hours | 0.013 (0.042) | -0.010 (0.093) | 0.018 (0.038) | -0.085 (0.036) | -0.107 (0.047)

5. Secondary Outcome: Change From Baseline in Serum Corrected Calcium
Time Frame: Baseline and 10 minutes, 30 minutes, 1 hour, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 36, 42 and 48 hours post-dose
Population: Modified intent-to-treat population with available data at each time point
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
mmol/L
  10 Minutes: number analyzed (Participants) | 7 | 6 | 6 | 6 | 6
  10 Minutes | -0.019 (0.047) | -0.008 (0.081) | -0.022 (0.063) | -0.017 (0.053) | -0.030 (0.049)
  30 Minutes | -0.018 (0.036) | -0.008 (0.079) | -0.018 (0.062) | -0.023 (0.041) | -0.042 (0.037)
  1 Hour | -0.024 (0.039) | -0.033 (0.073) | -0.023 (0.056) | -0.017 (0.058) | -0.042 (0.026)
  3 Hours: number analyzed (Participants) | 7 | 6 | 6 | 6 | 6
  3 Hours | -0.001 (0.035) | -0.002 (0.043) | -0.017 (0.048) | -0.025 (0.066) | -0.043 (0.028)
  6 Hours: number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
  6 Hours | -0.024 (0.040) | -0.048 (0.056) | 0.008 (0.066) | -0.045 (0.058) | -0.130 (0.069)
  9 Hours: number analyzed (Participants) | 8 | 5 | 6 | 5 | 6
  9 Hours | -0.010 (0.041) | -0.102 (0.079) | -0.120 (0.218) | -0.126 (0.043) | -0.163 (0.069)
  12 Hours | -0.032 (0.033) | -0.035 (0.048) | -0.067 (0.019) | -0.173 (0.026) | -0.228 (0.042)
  15 Hours | -0.154 (0.309) | -0.052 (0.072) | -0.107 (0.039) | -0.213 (0.064) | -0.255 (0.078)
  18 Hours | -0.067 (0.076) | -0.007 (0.063) | -0.100 (0.024) | -0.187 (0.058) | -0.272 (0.100)
  21 Hours: number analyzed (Participants) | 8 | 6 | 6 | 5 | 6
  21 Hours | -0.035 (0.040) | 0.012 (0.090) | -0.090 (0.023) | -0.150 (0.072) | -0.228 (0.056)
  24 Hours: number analyzed (Participants) | 8 | 6 | 6 | 5 | 5
  24 Hours | -0.015 (0.026) | -0.030 (0.048) | -0.018 (0.036) | -0.156 (0.031) | -0.214 (0.063)
  27 Hours | 0.040 (0.041) | 0.030 (0.085) | 0.038 (0.056) | -0.027 (0.050) | -0.115 (0.055)
  30 Hours: number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
  30 Hours | 0.008 (0.035) | 0.035 (0.078) | 0.007 (0.046) | -0.125 (0.067) | -0.138 (0.064)
  36 Hours | -0.025 (0.037) | 0.008 (0.046) | -0.038 (0.081) | -0.103 (0.068) | -0.157 (0.051)
  42 Hours: number analyzed (Participants) | 8 | 6 | 6 | 5 | 6
  42 Hours | 0.001 (0.060) | -0.023 (0.061) | 0.022 (0.026) | -0.056 (0.021) | -0.067 (0.036)
  48 Hours | 0.020 (0.033) | -0.007 (0.048) | 0.015 (0.022) | -0.048 (0.034) | -0.087 (0.030)

6. Secondary Outcome: Change From Baseline in Serum Phosphate
Time Frame: Baseline and 10 minutes, 30 minutes, 1 hour, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 36, 42 and 48 hours post-dose
Population: Modified intent-to-treat population with available data at each time point
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
mmol/L
  10 Minutes | -0.033 (0.035) | 0.007 (0.094) | -0.065 (0.059) | -0.010 (0.031) | 0.022 (0.042)
  30 Minutes | -0.041 (0.067) | -0.055 (0.085) | -0.067 (0.055) | -0.017 (0.042) | 0.012 (0.056)
  1 Hour | -0.055 (0.079) | -0.067 (0.124) | -0.058 (0.039) | -0.010 (0.045) | 0.005 (0.035)
  3 Hours: number analyzed (Participants) | 7 | 6 | 6 | 6 | 6
  3 Hours | 0.000 (0.093) | -0.013 (0.140) | 0.005 (0.096) | 0.110 (0.104) | 0.060 (0.083)
  6 Hours: number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
  6 Hours | 0.008 (0.153) | -0.088 (0.109) | 0.098 (0.123) | 0.058 (0.237) | 0.146 (0.142)
  9 Hours: number analyzed (Participants) | 8 | 5 | 6 | 5 | 6
  9 Hours | 0.130 (0.174) | 0.128 (0.122) | 0.100 (0.118) | 0.162 (0.135) | 0.275 (0.126)
  12 Hours | 0.015 (0.086) | 0.043 (0.123) | -0.090 (0.165) | -0.018 (0.164) | 0.028 (0.143)
  15 Hours | 0.228 (0.251) | 0.258 (0.132) | 0.188 (0.180) | 0.220 (0.139) | 0.355 (0.141)
  18 Hours | 0.381 (0.150) | 0.357 (0.120) | 0.307 (0.120) | 0.375 (0.113) | 0.538 (0.100)
  21 Hours: number analyzed (Participants) | 8 | 6 | 6 | 5 | 6
  21 Hours | 0.278 (0.164) | 0.315 (0.132) | 0.312 (0.065) | 0.296 (0.129) | 0.518 (0.120)
  24 Hours: number analyzed (Participants) | 8 | 6 | 6 | 5 | 5
  24 Hours | -0.003 (0.079) | 0.093 (0.099) | 0.053 (0.079) | 0.158 (0.126) | 0.116 (0.096)
  27 Hours | -0.085 (0.156) | -0.003 (0.124) | -0.127 (0.044) | -0.015 (0.215) | 0.065 (0.141)
  30 Hours: number analyzed (Participants) | 8 | 6 | 6 | 6 | 5
  30 Hours | 0.060 (0.210) | 0.085 (0.137) | 0.130 (0.157) | 0.148 (0.242) | 0.388 (0.087)
  36 Hours | 0.116 (0.127) | 0.162 (0.130) | 0.045 (0.082) | 0.072 (0.106) | 0.280 (0.210)
  42 Hours: number analyzed (Participants) | 8 | 6 | 6 | 5 | 6
  42 Hours | 0.335 (0.155) | 0.343 (0.123) | 0.342 (0.076) | 0.398 (0.222) | 0.480 (0.235)
  48 Hours | 0.044 (0.107) | 0.100 (0.087) | 0.027 (0.115) | 0.142 (0.162) | 0.160 (0.111)

7. Secondary Outcome: Percent Change From Baseline in Serum Calcitonin
Time Frame: Baseline and 10 minutes, 30 minutes, 3, 12, 24, and 48 hours post-dose
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
percent change
  10 Minutes | 15.92 (50.25) | 9.18 (14.47) | -5.07 (12.42) | 15.44 (29.09) | 51.45 (119.74)
  30 Minutes | 17.41 (57.12) | 16.72 (29.86) | 8.20 (37.05) | 24.39 (33.50) | 77.35 (143.22)
  3 Hours | 11.48 (25.51) | 3.33 (8.16) | -0.78 (17.80) | 3.12 (20.84) | 47.81 (109.64)
  12 Hours | 12.14 (52.58) | 10.56 (25.86) | -5.07 (12.42) | -10.89 (17.56) | 9.71 (28.64)
  24 Hours | 15.51 (61.10) | -1.11 (2.72) | -5.07 (12.42) | -13.45 (20.84) | -4.69 (11.48)
  48 Hours | 26.42 (74.89) | 5.00 (12.25) | -5.07 (12.42) | 0.53 (16.81) | 31.58 (88.51)

8. Secondary Outcome: Percent Change From Baseline in Serum 1,25 (OH)2 Vitamin D
Time Frame: Baseline and 12, 24, and 48 hours post-dose
Population: Modified intent-to-treat population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 8 | 6 | 6 | 6 | 6
percent change
  12 Hours | -14.46 (5.49) | -4.64 (12.06) | -6.12 (19.16) | -18.43 (9.44) | -25.60 (7.90)
  24 Hours | -0.61 (13.13) | 3.16 (16.23) | 4.16 (17.23) | -0.54 (15.12) | -14.51 (7.11)
  48 Hours | -4.32 (11.22) | 0.09 (19.03) | 5.99 (18.81) | 0.61 (11.49) | -3.53 (16.54)

9. Secondary Outcome: Maximum Observed Concentration (Cmax) for Etelcalcetide
Description: Plasma samples were analyzed for levels of etelcalcetide for pharmacokinetic (PK) analysis using a validated liquid chromatography/mass spectrometry (LC/MS) method.
Time Frame: Blood samples for PK assessment were drawn pre-dose, at 5, 10, 15, 20, and 30 minutes, post-dose, and at 1, 1.5, 2, 2.5, 3, 4, 6, 12, 24, 36, and 48 hours after drug administration.
Population: Participants who received etelcalcetide
Measure: Mean (Standard Deviation); unit: μg/L
Arm/Group | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
μg/L | 43.5 (7.86) | 171 (35.6) | 280 (59.3) | 583 (144)

10. Secondary Outcome: Area Under the Concentration-time Curve Between the Time of Dose and the Last Time Point (AUCall) for Etelcalcetide
Time Frame: as for outcome 9
Population: Participants who received etelcalcetide
Measure: Mean (Standard Deviation); unit: hr*μg/L
Arm/Group | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hr*μg/L | 81.1 (11.7) | 256 (32.5) | 544 (57.7) | 1130 (129)

11. Secondary Outcome: Observed Area Under the Concentration-time Curve Extrapolated to Infinity (AUCINFobs) for Etelcalcetide
Time Frame: as for outcome 9
Population: Participants who received etelcalcetide
Measure: Mean (Standard Deviation); unit: hr*μg/L
Arm/Group | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hr*μg/L | 94.3 (12.5) | 294 (34.1) | 623 (71.5) | 1290 (116)

12. Secondary Outcome: Percent Observed Area Under the Concentration-time Curve Extrapolated to Infinity Resulting From Extrapolation to Concentration of 0 ng/mL (AUC%Extrapobs)
Time Frame: as for outcome 9
Population: Participants who received etelcalcetide
Measure: Mean (Standard Deviation); unit: percentage of AUCINFobs
Arm/Group | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of AUCINFobs | 14.0 (1.33) | 13.2 (2.57) | 12.6 (2.43) | 12.0 (2.79)

13. Secondary Outcome: Terminal Elimination Rate Constant (λz) for Etelcalcetide
Time Frame: as for outcome 9
Population: Participants who received etelcalcetide
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
1/hr | 0.0357 (0.00246) | 0.0349 (0.00337) | 0.0378 (0.00486) | 0.0382 (0.00539)

14. Secondary Outcome: Half-life Associated With the Terminal (Log-linear) Elimination Phase (HLλz) for Etelcalcetide
Time Frame: as for outcome 9
Population: Participants who received etelcalcetide
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 19.5 (1.35) | 20.0 (2.25) | 18.6 (2.51) | 18.4 (2.21)

15. Secondary Outcome: Total Body Clearance (CL) for Etelcalcetide
Time Frame: as for outcome 9
Population: Participants who received etelcalcetide
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
L/hr | 5.38 (0.675) | 6.87 (0.750) | 8.11 (0.928) | 7.83 (0.755)

16. Secondary Outcome: Volume of Distribution at Steady State for Etelcalcetide
Time Frame: as for outcome 9
Population: Participants who received etelcalcetide
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
liters | 113 (19.6) | 138 (26.0) | 160 (21.0) | 152 (30.0)

17. Secondary Outcome: Number of Participants With Antibodies to Etelcalcetide
Description: Serum samples were analyzed for antibodies against etelcalcetide using a validated enzyme-linked immunosorbent assay (ELISA).
Time Frame: Samples for antibody analysis were collected pre-dose and between days 7-12 and days 21-28.
Population: Participants who received etelcalcetide
Measure: Count of Participants; unit: Participants
Arm/Group | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through 7 days
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Groups:
- Etelcalcetide Pooled: Participants received a single dose of etelcalcetide administered by intravenous injection.
Arm/Group | Pooled Placebo | Etelcalcetide 0.5 mg | Etelcalcetide 2 mg | Etelcalcetide 5 mg | Etelcalcetide 10 mg | Etelcalcetide Pooled
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6 | 0/6 | 0/6 | 0/6 | 0/24
Other Adverse Events (participants affected / at risk) | 2/8 | 0/6 | 1/6 | 2/6 | 2/6 | 5/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pooled Placebo (N=8) | Etelcalcetide 0.5 mg (N=6) | Etelcalcetide 2 mg (N=6) | Etelcalcetide 5 mg (N=6) | Etelcalcetide 10 mg (N=6) | Etelcalcetide Pooled (N=24)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
FEELING HOT (General disorders) | 0 | 0 | 1 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
LETHARGY (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.